CLINICAL TRIAL: NCT05116605
Title: Examining the Differential Effects of Photobiomodulation on Sleep and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2104299326
Record Dates: First submitted 2021-10-29; First posted 2021-11-11 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Sleep Quality
Keywords: Photobiomodulation; Sleep; Wearable Technology
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: All participants will complete the following design. Women who experience menstrual flow will be scheduled to ensure that flow occurs on weeks 4 & 8 for consistency.
  Baseline block (weeks 1-4): At intake, participants will complete up to 13 surveys, which includes 2 baseline questionnaires, & the first rendition of weekly & monthly surveys, as well as complete a physical performance task & 4 cognitive tasks. Participants will complete daily surveys each morning & night, & wear wearable devices to monitor physiology during sleep. A laboratory visit will occur once per week for completion of weekly surveys, as well as cognitive & physical performance assessments; monthly surveys will also be completed during the fourth week.
  Intervention block (weeks 5-8): Daily, weekly, & monthly activities described for the baseline block will continue; participants will additionally complete three 20-minute PBM sessions per week. The final week of this block will also involve an exit survey.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photobiomodulation (PBM) (Experimental): Participants will utilize the NovoTHOR whole body light pod
  Interventions: Other: Photobiomodulation (PBM)

INTERVENTIONS:
Other: Photobiomodulation (PBM) — Photobiomodulation (PBM) is light therapy in both the visible and near-infrared range (non-UV). This light is absorbed through the skin and functions at the cellular level, providing a lowering of inflammation and oxidative stress. Participants will undergo 20 minute sessions three times a week for 4 weeks using the NovoTHOR as the only intervention.
  Other Names: NovoTHOR Whole Body Light Bed

SUMMARY:
The objective of this research study is to assess how the implementation of photobiomodulation affects sleep quality, sleep structure, nocturnal physiology, subjective wellness, recovery from stressors, and resultant effects on performance and well-being.

DETAILED DESCRIPTION:
Photobiomodulation (PBM) is light therapy in both the visible and near-infrared range (non-UV). This light is absorbed through the skin and functions at the cellular level, providing a lowering of inflammation and oxidative stress. By provoking these photochemical changes, previous research indicates that PBM can provide both physical (e.g. pain reduction, strength enhancement) and cognitive benefits (e.g. increased memory extinction, improved cortical oxygen consumption). PBM is effective both preceding and succeeding functional tests, proving its ability to provide a preventative and rehabilitative impact on the functionality of cells and tissues. Metabolic changes to the cerebral cortex and the muscular system combine with anti-inflammatory and protective capabilities to augment recovery from physiological stressors. A plurality of literature reports light therapy given solely to specific body regions. However, partial body treatment may limit the comprehensive and systematic response to PBM treatment. Consequently, recent developments from commercial companies, such as NovoTHOR, have generated a consumer market for whole-body PBM. Yet, the physiological responses to these treatment modalities, as well as their effects on health and well-being is not fully understood.

Participants will undergo a four week block of baseline data collection, which involves nightly sleep monitoring, as well as daily, weekly, and monthly surveys and assessments. Following the baseline block, participants will complete a four week intervention block completing 3 PBM sessions per week. PBM sessions will be completed using the NovoThor light bed and will last 20 minutes in duration. Daily, weekly, and monthly monitoring and tasks will continue throughout this block.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-50 years of age

Exclusion Criteria:

* Has a head diameter outside the range of 20.8-24 inches, or an approved head-mounted EEG device doesn't otherwise fit properly
* Exceeds 290 pounds in body weight
* Has photophobia (light sensitivity)
* Has epilepsy or is prone to seizures
* Has thyroid problems or has been medicated for thyroid issues
* Has a current lower body musculoskeletal injury
* Has a current injury requiring an irremovable cast
* Is pregnant or actively trying to become pregnant
* Has a known or diagnosed sleep disorder
* Females who have become menopausal or are exhibiting signs or symptoms of becoming perimenopausal
* Females who are unable to identify when their monthly menstrual period will occur
* Individuals who work during the night shift or have significantly abnormal sleep schedule
* Has undergone travel across more than two collective time zones in the last two weeks
* Individuals who intend to have any significant medical procedures scheduled to occur within 12 weeks of enrollment
* Individuals who have intentions, or have discussed with their doctor, about adding or making any alterations to their prescribed medications within 12 weeks of enrollment
* Individuals who have any travel plans or other obligations within 12 weeks of enrollment that would prevent them from completing study requirements and attending required laboratory visits
* Individuals who intend to make significant alterations to their sleeping patterns within 12 weeks of enrollment. This may include, but is not limited to, changes such as moving, getting a new mattress, having someone move in with them, etc.
* Does not meet the ACSM's guidelines for exercise prescription. This is defined as:

  1. Presenting with an absolute contraindication OR

     1. Has a known cardiovascular, pulmonary, renal, metabolic disease, or other chronic illness
     2. Presents with symptoms indicating cardiovascular, pulmonary, renal, or metabolic disease
  2. presenting with two or more relative contraindications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Change in Nocturnal Heart Rate as measured by OURA Ring | Daily from baseline through study completion at 8 weeks
  Heart rate (beats per minute) will be quantified throughout the night via the OURA ring.
Change in Subjective Sleep Quality | Daily from baseline through study completion at 8 weeks
  A custom daily morning questionnaire will be used to record how a participant feels the quality of their sleep was the previous night (e.g. 1, very poor; 10 excellent). This questionnaire will be taken on the participants smartphone within 30 minutes of waking.
Change in Nocturnal Heart Rate Variability as measured by OURA Ring | Daily from baseline through study completion at 8 weeks
  Heart rate variability will be quantified throughout the night via the OURA ring.
Subjective Success of PBM assessed via Survey | Once at the end of week 8
  Following completion of the study, a custom questionnaire will record how successful the participant believes PBM was in improving their sleep and well being.
Changes in Subjective Anxiety as measured via the STAI | Monthly from baseline through study completion at 8 weeks
  Participants will complete the previously validated State Trait Anxiety Index (STAI) as a measure of subjective anxiety, where higher scores are suggestive of greater anxiety.
Changes in Subjective Sleep as measured via PSQI | Monthly from baseline through study completion at 8 weeks
  Participant's subjective reports of sleep quality will be quantified through the previously validated Pittsburgh Sleep Quality Index (PSQI). Questions are scored into multiple components to determine sleep difficulty in various areas, where higher scores are indicative of greater sleep difficulties; these scores will be compared across timepoints.
Changes in Perceived Stress as measured via PSS | Weekly from baseline through study completion at 8 weeks
  Participants' perceived stress will be quantified via the previously validated Perceived Stress Scale (PSS), which asks participants to report on the frequency of various experiences (0, never; 4, very often) and final scoring suggests lower scores to be associated with lower levels of stress.
Change in Subjective Epworth Sleepiness Scale measured via questionnaire | Weekly throughout study completion at 8 weeks
  Participants will complete previously validated questionnaires as often as weekly.
  Epworth Sleepiness Scale (ESS) - eight-item questionnaire assessing sleep behaviors on a scale of 0 to 3. Higher scores = increased average sleep propensity in daily life
Change in Eriksen Flanker Task | Changes from baseline versus end of study week 8
  The Flanker Task is a response inhibition test used to assess the participant's ability to suppress a response that is inappropriate based on the task rules. Participants are to respond, left or right, to the direction of the middle arrow (target arrow) of five aligned items. The task consists of congruent stimulus (the direction of the target arrow and flanker arrows are the same), incongruent stimulus (the direction of the target arrow is opposite of the flanker arrows), and neutral stimulus (flanker items are different then the target arrow). The dependent variable is the measurement of reaction time to select the direction of the target arrow.
Change in Psychomotor Vigilance Task | Changes from baseline versus end of study week 8
  A reaction time test that measures a person's sustained attention to a cue presented on a screen at random inter-stimulus intervals. In addition to the measures of reaction time to correct responses the errors of commission (responding when there is not response cue) and omission (failing to respond to a response cue).

SECONDARY OUTCOMES:
Change in Subjective Restorative Sleep Questionnaire | Weekly throughout study completion at 8 weeks
  Participants will complete previously validated questionnaires as often as weekly.
  Restorative Sleep Questionnaire (RSQ) - nine-item questionnaire assessing sleep behaviors on a scale of 0 to 5. Higher scores = better sleep
Changes in Sleep Disturbances as measured via the Sleep Disorders Questionnaire | Monthly from baseline through study completion at 8 weeks
  Participants will complete a 34 item checklist that has been previously used for screening of a potential sleep disorder; the more items that the participant feels applies to them, the higher the likelihood of the individual having a sleep disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Rockefeller Neuroscience Institute at West Virginia University, Morgantown, West Virginia, United States